CLINICAL TRIAL: NCT00982696
Title: Treatment of Advanced Head and Neck Cancer With Opioid Growth Factors: Phase II
Brief Title: Treatment of Advanced Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Deemed ineffective
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, David Goldenberg, Associate Professor of Medicine and Surgery, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSU 23429; NCT00905099 (obsolete NCT alias)
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
Keywords: head and neck cancer; opioid growth factor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Enkephalin, Methionine; Opioid Peptides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Opioid Growth Factor (OGF)
  Interventions: Biological: Opioid Growth Factor

INTERVENTIONS:
Biological: Opioid Growth Factor — 250ug per kilogram weekly IV infusions
  Other Names: endogenous opioid peptide; Met-enkephalin

SUMMARY:
This study will investigate the efficacy of opioid growth factor (OGF) on tumor size and survival in patients with head and neck cancer who have failed standard therapy.

DETAILED DESCRIPTION:
The major focus of the study will involve assessment of tumor response, patient survival, tolerance to drug, quality of life, depression, pain management and nutrition. During the study we will begin to study the kinetics of opioid growth factor (OGF) exogenous administration and the relationship between plasma OGF levels, stage of disease and length of treatment. Apart from potentially having growth inhibitory action on cancer, OGF may have some psychological and other biological effects which may prove to be beneficial in the patient's treatment. Presently there is no effective therapy or quality of life adjuvants for the 30,000 Americans who develop head and neck cancer yearly.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and cytologically confirmed diagnosis of squamous cell carcinoma.
* Patients not amenable to curative treatments with further surgery and/or radiation.
* Patient has failed treatment with chemotherapy
* Lesions must be distinct and the minimum measurements must be at least 2.0 cm x 2.0 cm at baseline.
* Karnofsky performance rating of at lest 50%.

Exclusion Criteria:

* Patients with severe and unstable cardiovascular disease.
* Treatment naive subjects will not be included for study.
* Patients with poorly controlled diabetes, seizure disorder, primary CNS tumors or known brain metastases will be excluded.
* Pregnant or nursing women.
* Patients requiring antibiotics in the preceding 2 weeks for a serious infection are not eligible.
* Patients with a fever > 37.8 degrees C.
* Pulse < 60 or > 110
* Systolic blood pressure > 170 or less than 90 are not eligible.
* Patients with nasopharyngeal squamous cell carcinoma will be excluded
* Patients with hypercalcemia will be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Progression of tumor measured with CT scan | every 3 months

SECONDARY OUTCOMES:
Metastatic development using CT scan | every 3 months

OTHER OUTCOMES:
Pharmacokinetics of OGF | every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Goldenberg, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Zagon IS, McLaughlin PJ. Endogenous opioid systems regulate growth of neural tumor cells in culture. Brain Res. 1989 Jun 19;490(1):14-25. doi: 10.1016/0006-8993(89)90425-3. PMID 2758319
- [Background] Wybran J, Schandene L, Van Vooren JP, Vandermoten G, Latinne D, Sonnet J, De Bruyere M, Taelman H, Plotnikoff NP. Immunologic properties of methionine-enkephalin, and therapeutic implications in AIDS, ARC, and cancer. Ann N Y Acad Sci. 1987;496:108-14. doi: 10.1111/j.1749-6632.1987.tb35753.x. No abstract available. PMID 3496822
- [Background] Zagon IS, McLaughlin PJ. Opioid antagonists inhibit the growth of metastatic murine neuroblastoma. Cancer Lett. 1983 Nov;21(1):89-94. doi: 10.1016/0304-3835(83)90087-3. PMID 6640516
- [Background] Goldenberg D, Zagon IS, Fedok F, Crist HS, McLaughlin PJ. Expression of opioid growth factor (OGF)-OGF receptor (OGFr) axis in human nonmedullary thyroid cancer. Thyroid. 2008 Nov;18(11):1165-70. doi: 10.1089/thy.2008.0112. PMID 19014324
- See also: Penn State Hershey Cancer Institute — http://www.pennstatehershey.org/web/cancer/research